CLINICAL TRIAL: NCT03254420
Title: Randomized Phase II Study Evaluating Late Toxicity Following Intensity-Modulated Radiotherapy and Two Image-Guided Strategies With Corresponding Treatment Margins. (RCMIGI)
Brief Title: Evaluation of Late Toxicity Following Intensity-Modulated Radiotherapy and Two Image-Guided Strategies With Corresponding Treatment Margins.
Acronym: RCMIGI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICM-URC2015/33
Record Dates: First submitted 2017-08-16; First posted 2017-08-18 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Image-guided radiation therapy (IGRT) with standard margins (Active Comparator): moderate hypofractionation during 4 weeks
  Interventions: Radiation: moderate hypofractionation Radiotherapy
- Calypso tracking system with margin reduction (Experimental): moderate hypofractionation during 4 weeks after calypso beacon implant 10 days before
  Interventions: Device: Calypso beacon implant; Radiation: moderate hypofractionation Radiotherapy

INTERVENTIONS:
Device: Calypso beacon implant — Calypso beacon implant before radiotherapy
  Arms: Calypso tracking system with margin reduction
Radiation: moderate hypofractionation Radiotherapy — moderate hypofractionation Radiotherapy

SUMMARY:
The Calypso® System (Varian Medical Systems, Inc., Palo Alto, CA) is a recent technology using electromagnetic transponders implanted within the prostate. It is a real-time target tracking system that takes into account both inter- and intrafractional target motion. So the exact position and movement of the prostate can be determined during radiation therapy treatment.

The aim of this study is to assess pelvic late toxicity rate after intensity-modulated radiotherapy (IMRT) when using the Calypso® System with a reduction of treatment margins. In this randomized study, patients will receive IGRT treatment using the Calypso system or a conventional IGRT treatment.

DETAILED DESCRIPTION:
Prostate cancer is the most frequent cancer in men. Radiotherapy is one of the reference treatments for localized prostate cancer. Prostate was initially thought to be a non-moving target, but the newest reports have raised the contrary as evidence. Image-guided radiotherapy (IGRT) is a current standard treatment for localized prostate cancer which enables to take into account interfractional prostate motion before treatment.

The Calypso® System (Varian Medical Systems, Inc., Palo Alto, CA) is a recent technology using electromagnetic transponders implanted within the prostate. It is a real-time target tracking system that takes into account both inter- and intrafractional target motion. So the exact position and movement of the prostate can be determined during radiation therapy treatment.

As Planned Target Volume (PTV) margins integrate set-up margins and the management of organ motion, margin reduction can reasonably be considered in case of target motion management improvement.

To date, no prospective randomized clinical data is available using this technique for the treatment of low- or intermediate-risk prostate cancer patients with modern standard fractionation radiotherapy and image guidance.

The aim of this study is to assess pelvic late toxicity rate after intensity-modulated radiotherapy (IMRT) when using the Calypso® System with a reduction of treatment margins. In this randomized study, patients will receive IGRT treatment using the Calypso system or a conventional IGRT treatment.

ELIGIBILITY:
Inclusion Criteria:

* Localized prostate cancer, histologically proven.
* No evidence of metastases (M0). No evidence of lymph nodes involvement (N0) (bilateral lymph node dissection is not mandatory if lymph node involvement risk is low according to the Partin tables).
* Low-risk or intermediate clinical stage according to the D'Amico classification (T1-T2 and Gleason < 8 and PSA < 20 ng/ml) (appendix 3).
* No grade > 2 urinary or rectal clinical sign or symptom according to the CTCAE V4.03 scale.
* Performance status ECOG ≤ 1.
* No hip prosthesis or metallic vascular graft near the prostate.
* No endopenian stent.
* No pace maker, implanted defibrillator or neurostimulator.
* No allergy to local anesthetics.
* No irreversible anticoagulation or antiplatelet treatment for the implantation period.
* Pelvic and abdominal anatomy compatible with the use of the Calypso® system (predictive detector to fiducials distance less than 19 cm, evaluated on planning CT-scan) (distance from skin surface to prostate center less than 17 cm).
* Patient aged ≥ 18 and less than 80 years old.
* Dated and signed written informed consent available.
* Patients must be affiliated to a French Social Security System.

Exclusion Criteria:

* Indication of pelvic nodes irradiation.
* Prior pelvic irradiation.
* Biopsy-proven seminal vesicle invasion.
* Prior bilateral orchiectomy.
* Prior radical prostatectomy.
* Other malignancy except adequately-treated basal cell carcinoma of the skin or other malignancy from which the patient has been disease-free for at least 5 years.
* Psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
* Other uncontrolled systemic disease (cardiovascular, renal, liver, pulmonary embolism, etc.).
* Known VIH positive patients (no specific test needed).
* Known homozygote ATM Mutation (Ataxia telengiectasia).

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2028-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Riou Olivier, Study Chair — Institut régional du Cancer de Montpellier
Locations (1):
- Institut regional du Cancer - Val d Aurelle, Montpellier, France

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients

REFERENCES:
- [Background] Jereczek-Fossa BA, Orecchia R. Evidence-based radiation oncology: definitive, adjuvant and salvage radiotherapy for non-metastatic prostate cancer. Radiother Oncol. 2007 Aug;84(2):197-215. doi: 10.1016/j.radonc.2007.04.013. Epub 2007 May 29. PMID 17532494
- [Background] Zaorsky NG, Harrison AS, Trabulsi EJ, Gomella LG, Showalter TN, Hurwitz MD, Dicker AP, Den RB. Evolution of advanced technologies in prostate cancer radiotherapy. Nat Rev Urol. 2013 Oct;10(10):565-79. doi: 10.1038/nrurol.2013.185. Epub 2013 Sep 10. PMID 24018567
- [Background] Budaus L, Bolla M, Bossi A, Cozzarini C, Crook J, Widmark A, Wiegel T. Functional outcomes and complications following radiation therapy for prostate cancer: a critical analysis of the literature. Eur Urol. 2012 Jan;61(1):112-27. doi: 10.1016/j.eururo.2011.09.027. Epub 2011 Oct 6. PMID 22001105
- [Background] Ohri N, Dicker AP, Showalter TN. Late toxicity rates following definitive radiotherapy for prostate cancer. Can J Urol. 2012 Aug;19(4):6373-80. PMID 22892261
- [Background] Pardo Y, Guedea F, Aguilo F, Fernandez P, Macias V, Marino A, Hervas A, Herruzo I, Ortiz MJ, Ponce de Leon J, Craven-Bratle J, Suarez JF, Boladeras A, Pont A, Ayala A, Sancho G, Martinez E, Alonso J, Ferrer M. Quality-of-life impact of primary treatments for localized prostate cancer in patients without hormonal treatment. J Clin Oncol. 2010 Nov 1;28(31):4687-96. doi: 10.1200/JCO.2009.25.3245. Epub 2010 Oct 4. PMID 20921463
- [Background] de Crevoisier R, Fiorino C, Dubray B. [Dosimetric factors predictive of late toxicity in prostate cancer radiotherapy]. Cancer Radiother. 2010 Oct;14(6-7):460-8. doi: 10.1016/j.canrad.2010.07.225. Epub 2010 Aug 24. French. PMID 20797890
- [Background] Valdagni R, Rancati T, Fiorino C. Predictive models of toxicity with external radiotherapy for prostate cancer: clinical issues. Cancer. 2009 Jul 1;115(13 Suppl):3141-9. doi: 10.1002/cncr.24356. PMID 19544543
- [Background] Yu JB. Hypofractionated Radiotherapy for Prostate Cancer: Further Evidence to Tip the Scales. J Clin Oncol. 2017 Jun 10;35(17):1867-1869. doi: 10.1200/JCO.2017.72.7016. Epub 2017 Mar 29. No abstract available. PMID 28355114
- [Background] Dearnaley D, Syndikus I, Mossop H, Khoo V, Birtle A, Bloomfield D, Graham J, Kirkbride P, Logue J, Malik Z, Money-Kyrle J, O'Sullivan JM, Panades M, Parker C, Patterson H, Scrase C, Staffurth J, Stockdale A, Tremlett J, Bidmead M, Mayles H, Naismith O, South C, Gao A, Cruickshank C, Hassan S, Pugh J, Griffin C, Hall E; CHHiP Investigators. Conventional versus hypofractionated high-dose intensity-modulated radiotherapy for prostate cancer: 5-year outcomes of the randomised, non-inferiority, phase 3 CHHiP trial. Lancet Oncol. 2016 Aug;17(8):1047-1060. doi: 10.1016/S1470-2045(16)30102-4. Epub 2016 Jun 20. PMID 27339115
- [Background] Lee WR, Dignam JJ, Amin MB, Bruner DW, Low D, Swanson GP, Shah AB, D'Souza DP, Michalski JM, Dayes IS, Seaward SA, Hall WA, Nguyen PL, Pisansky TM, Faria SL, Chen Y, Koontz BF, Paulus R, Sandler HM. Randomized Phase III Noninferiority Study Comparing Two Radiotherapy Fractionation Schedules in Patients With Low-Risk Prostate Cancer. J Clin Oncol. 2016 Jul 10;34(20):2325-32. doi: 10.1200/JCO.2016.67.0448. Epub 2016 Apr 4. PMID 27044935
- [Background] Incrocci L, Wortel RC, Alemayehu WG, Aluwini S, Schimmel E, Krol S, van der Toorn PP, Jager H, Heemsbergen W, Heijmen B, Pos F. Hypofractionated versus conventionally fractionated radiotherapy for patients with localised prostate cancer (HYPRO): final efficacy results from a randomised, multicentre, open-label, phase 3 trial. Lancet Oncol. 2016 Aug;17(8):1061-1069. doi: 10.1016/S1470-2045(16)30070-5. Epub 2016 Jun 20. PMID 27339116
- [Background] Arcangeli G, Saracino B, Arcangeli S, Gomellini S, Petrongari MG, Sanguineti G, Strigari L. Moderate Hypofractionation in High-Risk, Organ-Confined Prostate Cancer: Final Results of a Phase III Randomized Trial. J Clin Oncol. 2017 Jun 10;35(17):1891-1897. doi: 10.1200/JCO.2016.70.4189. Epub 2017 Mar 29. PMID 28355113
- [Background] Catton CN, Lukka H, Gu CS, Martin JM, Supiot S, Chung PWM, Bauman GS, Bahary JP, Ahmed S, Cheung P, Tai KH, Wu JS, Parliament MB, Tsakiridis T, Corbett TB, Tang C, Dayes IS, Warde P, Craig TK, Julian JA, Levine MN. Randomized Trial of a Hypofractionated Radiation Regimen for the Treatment of Localized Prostate Cancer. J Clin Oncol. 2017 Jun 10;35(17):1884-1890. doi: 10.1200/JCO.2016.71.7397. Epub 2017 Mar 15. PMID 28296582
- [Background] Mottet N, van den Bergh RCN, Briers E, Van den Broeck T, Cumberbatch MG, De Santis M, Fanti S, Fossati N, Gandaglia G, Gillessen S, Grivas N, Grummet J, Henry AM, van der Kwast TH, Lam TB, Lardas M, Liew M, Mason MD, Moris L, Oprea-Lager DE, van der Poel HG, Rouviere O, Schoots IG, Tilki D, Wiegel T, Willemse PM, Cornford P. EAU-EANM-ESTRO-ESUR-SIOG Guidelines on Prostate Cancer-2020 Update. Part 1: Screening, Diagnosis, and Local Treatment with Curative Intent. Eur Urol. 2021 Feb;79(2):243-262. doi: 10.1016/j.eururo.2020.09.042. Epub 2020 Nov 7. PMID 33172724
- [Background] Rodin D, Tawk B, Mohamad O, Grover S, Moraes FY, Yap ML, Zubizarreta E, Lievens Y. Hypofractionated radiotherapy in the real-world setting: An international ESTRO-GIRO survey. Radiother Oncol. 2021 Apr;157:32-39. doi: 10.1016/j.radonc.2021.01.003. Epub 2021 Jan 14. PMID 33453312
- [Background] Chapet O, Decullier E, Bin S, Faix A, Ruffion A, Jalade P, Fenoglietto P, Udrescu C, Enachescu C, Azria D. Prostate hypofractionated radiation therapy with injection of hyaluronic acid: acute toxicities in a phase 2 study. Int J Radiat Oncol Biol Phys. 2015 Mar 15;91(4):730-6. doi: 10.1016/j.ijrobp.2014.11.027. PMID 25752385
- [Background] Palombarini M, Mengoli S, Fantazzini P, Cadioli C, Degli Esposti C, Frezza GP. Analysis of inter-fraction setup errors and organ motion by daily kilovoltage cone beam computed tomography in intensity modulated radiotherapy of prostate cancer. Radiat Oncol. 2012 Apr 2;7:56. doi: 10.1186/1748-717X-7-56. PMID 22472040
- [Background] Tanyi JA, He T, Summers PA, Mburu RG, Kato CM, Rhodes SM, Hung AY, Fuss M. Assessment of planning target volume margins for intensity-modulated radiotherapy of the prostate gland: role of daily inter- and intrafraction motion. Int J Radiat Oncol Biol Phys. 2010 Dec 1;78(5):1579-85. doi: 10.1016/j.ijrobp.2010.02.001. Epub 2010 May 14. PMID 20472357
- [Background] Nguyen NP, Davis R, Bose SR, Dutta S, Vinh-Hung V, Chi A, Godinez J, Desai A, Woods W, Altdorfer G, D'Andrea M, Karlsson U, Vo RA, Sroka T; International Geriatric Radiotherapy Group. Potential applications of image-guided radiotherapy for radiation dose escalation in patients with early stage high-risk prostate cancer. Front Oncol. 2015 Feb 2;5:18. doi: 10.3389/fonc.2015.00018. eCollection 2015. PMID 25699239
- [Background] Crehange G, Martin E, Supiot S, Chapet O, Mazoyer F, Naudy S, Maingon P. [Image-guided radiotherapy in prostate cancer: concepts and implications]. Cancer Radiother. 2012 Sep;16(5-6):430-8. doi: 10.1016/j.canrad.2012.07.183. Epub 2012 Aug 23. French. PMID 22921961
- [Background] Bernchou U, Agergaard SN, Brink C. Radiopaque marker motion during pre-treatment CBCT as a predictor of intra-fractional prostate movement. Acta Oncol. 2013 Aug;52(6):1168-74. doi: 10.3109/0284186X.2012.747698. Epub 2012 Dec 17. PMID 23244674
- [Background] Badakhshi H, Wust P, Budach V, Graf R. Image-guided radiotherapy with implanted markers and kilovoltage imaging and 6-dimensional position corrections for intrafractional motion of the prostate. Anticancer Res. 2013 Sep;33(9):4117-21. PMID 24023358
- [Background] Tong X, Chen X, Li J, Xu Q, Lin MH, Chen L, Price RA, Ma CM. Intrafractional prostate motion during external beam radiotherapy monitored by a real-time target localization system. J Appl Clin Med Phys. 2015 Mar 8;16(2):5013. doi: 10.1120/jacmp.v16i2.5013. PMID 26103174
- [Background] Das S, Liu T, Jani AB, Rossi P, Shelton J, Shi Z, Khan MK. Comparison of image-guided radiotherapy technologies for prostate cancer. Am J Clin Oncol. 2014 Dec;37(6):616-23. doi: 10.1097/COC.0b013e31827e4eb9. PMID 23428948
- [Background] Foster RD, Pistenmaa DA, Solberg TD. A comparison of radiographic techniques and electromagnetic transponders for localization of the prostate. Radiat Oncol. 2012 Jun 21;7:101. doi: 10.1186/1748-717X-7-101. PMID 22720845
- [Background] Korreman S, Rasch C, McNair H, Verellen D, Oelfke U, Maingon P, Mijnheer B, Khoo V. The European Society of Therapeutic Radiology and Oncology-European Institute of Radiotherapy (ESTRO-EIR) report on 3D CT-based in-room image guidance systems: a practical and technical review and guide. Radiother Oncol. 2010 Feb;94(2):129-44. doi: 10.1016/j.radonc.2010.01.004. Epub 2010 Feb 12. PMID 20153908
- [Background] Santanam L, Malinowski K, Hubenshmidt J, Dimmer S, Mayse ML, Bradley J, Chaudhari A, Lechleiter K, Goddu SK, Esthappan J, Mutic S, Low DA, Parikh P. Fiducial-based translational localization accuracy of electromagnetic tracking system and on-board kilovoltage imaging system. Int J Radiat Oncol Biol Phys. 2008 Mar 1;70(3):892-9. doi: 10.1016/j.ijrobp.2007.10.005. PMID 18262100
- [Background] Langen KM, Willoughby TR, Meeks SL, Santhanam A, Cunningham A, Levine L, Kupelian PA. Observations on real-time prostate gland motion using electromagnetic tracking. Int J Radiat Oncol Biol Phys. 2008 Jul 15;71(4):1084-90. doi: 10.1016/j.ijrobp.2007.11.054. Epub 2008 Feb 14. PMID 18280057
- [Background] Willoughby TR, Kupelian PA, Pouliot J, Shinohara K, Aubin M, Roach M 3rd, Skrumeda LL, Balter JM, Litzenberg DW, Hadley SW, Wei JT, Sandler HM. Target localization and real-time tracking using the Calypso 4D localization system in patients with localized prostate cancer. Int J Radiat Oncol Biol Phys. 2006 Jun 1;65(2):528-34. doi: 10.1016/j.ijrobp.2006.01.050. PMID 16690435
- [Background] Mayyas E, Chetty IJ, Chetvertkov M, Wen N, Neicu T, Nurushev T, Ren L, Lu M, Stricker H, Pradhan D, Movsas B, Elshaikh MA. Evaluation of multiple image-based modalities for image-guided radiation therapy (IGRT) of prostate carcinoma: a prospective study. Med Phys. 2013 Apr;40(4):041707. doi: 10.1118/1.4794502. PMID 23556877
- [Background] Noel C, Parikh PJ, Roy M, Kupelian P, Mahadevan A, Weinstein G, Enke C, Flores N, Beyer D, Levine L. Prediction of intrafraction prostate motion: accuracy of pre- and post-treatment imaging and intermittent imaging. Int J Radiat Oncol Biol Phys. 2009 Mar 1;73(3):692-8. doi: 10.1016/j.ijrobp.2008.04.076. Epub 2008 Aug 7. PMID 18692324
- [Background] Zhu M, Bharat S, Michalski JM, Gay HA, Hou WH, Parikh PJ. Adaptive radiation therapy for postprostatectomy patients using real-time electromagnetic target motion tracking during external beam radiation therapy. Int J Radiat Oncol Biol Phys. 2013 Mar 15;85(4):1038-44. doi: 10.1016/j.ijrobp.2012.08.001. Epub 2012 Sep 25. PMID 23021439
- [Background] Su Z, Zhang L, Murphy M, Williamson J. Analysis of prostate patient setup and tracking data: potential intervention strategies. Int J Radiat Oncol Biol Phys. 2011 Nov 1;81(3):880-7. doi: 10.1016/j.ijrobp.2010.07.1978. Epub 2010 Oct 8. PMID 20934274
- [Background] Kupelian P, Willoughby T, Mahadevan A, Djemil T, Weinstein G, Jani S, Enke C, Solberg T, Flores N, Liu D, Beyer D, Levine L. Multi-institutional clinical experience with the Calypso System in localization and continuous, real-time monitoring of the prostate gland during external radiotherapy. Int J Radiat Oncol Biol Phys. 2007 Mar 15;67(4):1088-98. doi: 10.1016/j.ijrobp.2006.10.026. Epub 2006 Dec 21. PMID 17187940
- [Background] Klayton T, Price R, Buyyounouski MK, Sobczak M, Greenberg R, Li J, Keller L, Sopka D, Kutikov A, Horwitz EM. Prostate bed motion during intensity-modulated radiotherapy treatment. Int J Radiat Oncol Biol Phys. 2012 Sep 1;84(1):130-6. doi: 10.1016/j.ijrobp.2011.11.041. Epub 2012 Feb 11. PMID 22330987
- [Background] Mantz C. A Phase II Trial of Stereotactic Ablative Body Radiotherapy for Low-Risk Prostate Cancer Using a Non-Robotic Linear Accelerator and Real-Time Target Tracking: Report of Toxicity, Quality of Life, and Disease Control Outcomes with 5-Year Minimum Follow-Up. Front Oncol. 2014 Nov 14;4:279. doi: 10.3389/fonc.2014.00279. eCollection 2014. PMID 25452933
- [Background] Sandler HM, Liu PY, Dunn RL, Khan DC, Tropper SE, Sanda MG, Mantz CA. Reduction in patient-reported acute morbidity in prostate cancer patients treated with 81-Gy Intensity-modulated radiotherapy using reduced planning target volume margins and electromagnetic tracking: assessing the impact of margin reduction study. Urology. 2010 May;75(5):1004-8. doi: 10.1016/j.urology.2009.10.072. Epub 2010 Feb 13. PMID 20153881
- [Background] Ozsahin M, Crompton NE, Gourgou S, Kramar A, Li L, Shi Y, Sozzi WJ, Zouhair A, Mirimanoff RO, Azria D. CD4 and CD8 T-lymphocyte apoptosis can predict radiation-induced late toxicity: a prospective study in 399 patients. Clin Cancer Res. 2005 Oct 15;11(20):7426-33. doi: 10.1158/1078-0432.CCR-04-2634. PMID 16243816
- [Background] Azria D, Betz M, Bourgier C, Jeanneret Sozzi W, Ozsahin M. Identifying patients at risk for late radiation-induced toxicity. Crit Rev Oncol Hematol. 2012 Dec;84 Suppl 1:e35-41. doi: 10.1016/j.critrevonc.2010.08.003. Epub 2010 Sep 24. PMID 20869261
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Rosen RC, Riley A, Wagner G, Osterloh IH, Kirkpatrick J, Mishra A. The international index of erectile function (IIEF): a multidimensional scale for assessment of erectile dysfunction. Urology. 1997 Jun;49(6):822-30. doi: 10.1016/s0090-4295(97)00238-0. PMID 9187685
- [Background] Nyaga VN, Arbyn M, Aerts M. Metaprop: a Stata command to perform meta-analysis of binomial data. Arch Public Health. 2014 Nov 10;72(1):39. doi: 10.1186/2049-3258-72-39. eCollection 2014. PMID 25810908

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Image-guided Radiation Therapy (IGRT) With Standard Margins | Calypso Tracking System With Margin Reduction
Started | 29 | 45
Completed | 26 | 44
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Image-guided Radiation Therapy (IGRT) With Standard Margins | Calypso Tracking System With Margin Reduction | Total
Number analyzed (Participants) | 29 | 45 | 74
Age, Continuous [Mean (Full Range); unit: years] | 68 [52 to 78] | 70 [51 to 78] | 69.5 [51 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 29 | 45 | 74
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Grade > 2 Late Pelvic Toxicities
Description: assessment of grade > 2 late pelvic toxicities between 3 months and 2 years after radiation period
Time Frame: between 3 months and 2 years after radiation period
Population: failure : presence of grade > 2 late pelvic toxicities between 3 months and 2 years after radiation period success : absence of grade > 2 late pelvic toxicities between 3 months and 2 years after radiation period
Measure: Count of Participants; unit: Participants
Arm/Group | Image-guided Radiation Therapy (IGRT) With Standard Margins | Calypso Tracking System With Margin Reduction
Number analyzed (Participants) | 26 | 44
Participants
  failure | 5 | 5
  success | 21 | 39

2. Secondary Outcome: Biological Relapse-free Survival
Description: evaluate at 5 years with PSA dosage
Time Frame: at 5 years after the radiotherapy
Measure: Number; unit: participants
Arm/Group | Image-guided Radiation Therapy (IGRT) With Standard Margins | Calypso Tracking System With Margin Reduction
Number analyzed (Participants) | 26 | 44
participants | 26 | 37

3. Secondary Outcome: Uncomplicated Survival (Local Recurrence or Metastatic Recurrence)
Description: evaluate et 5 years after the treatment with radiological exam
Time Frame: at 5 years after the radiotherapy
Measure: Number; unit: participants
Arm/Group | Image-guided Radiation Therapy (IGRT) With Standard Margins | Calypso Tracking System With Margin Reduction
Number analyzed (Participants) | 26 | 44
participants | 26 | 41

4. Secondary Outcome: Overall Survival
Description: number of death from baseline to 5 years after the treatment
Time Frame: from the baseline to 5 years after the radiotherapy
Measure: Number; unit: participants
Arm/Group | Image-guided Radiation Therapy (IGRT) With Standard Margins | Calypso Tracking System With Margin Reduction
Number analyzed (Participants) | 26 | 44
participants | 0 | 2

ADVERSE EVENTS:
Time Frame: adverse event data were collected from the baseline to 5 years after the radiotherapy
Arm/Group | Image-guided Radiation Therapy (IGRT) With Standard Margins | Calypso Tracking System With Margin Reduction
All-Cause Mortality (participants affected / at risk) | 0/26 | 2/44
Serious Adverse Events (participants affected / at risk) | 2/26 | 9/44
Other Adverse Events (participants affected / at risk) | 26/26 | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Image-guided Radiation Therapy (IGRT) With Standard Margins (N=26) | Calypso Tracking System With Margin Reduction (N=44)
hemovhromatosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
lithiasis choledocholithiasis grade 3 (Hepatobiliary disorders) | 1 (1) | 0 (0)
prostatitis grade 3 (Reproductive system and breast disorders) | 0 (0) | 2 (2)
thrombocytopenia grade 4 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
basela cell carcinoma grade 2 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
vascular stent stenosis grade 3 (General disorders) | 0 (0) | 1 (1)
peripheral artery stenosis grade 3 (Vascular disorders) | 0 (0) | 1 (1)
malignant melanoma grade 2 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
colon cancer metastatic grade 5 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
cerebral hematoma grade 3 (Nervous system disorders) | 0 (0) | 1 (1)
large instestine polyp grade 2 (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Image-guided Radiation Therapy (IGRT) With Standard Margins (N=26) | Calypso Tracking System With Margin Reduction (N=44)
blood and lymphatic (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — grade 4
ocular infection (Eye disorders) | 1 (1) | 0 (0) — grade 1
gastrointestinal disorders (Gastrointestinal disorders) | 16 (16) | 28 (28) — grade 1 and 2
general disorders and reaction at the site of administration (General disorders) | 10 (10) | 13 (13) — grade 1 and 2
Infections and infestations (Infections and infestations) | 0 (0) | 1 (1) — grade 2
hepatobiliary disorders (Hepatobiliary disorders) | 1 (1) | 0 (0) — grade 3
investigations (Investigations) | 1 (1) | 1 (1) — grade 1
musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) — grade 1 and 2
nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1) — grade 1
psychiatric disorders (Psychiatric disorders) | 6 (6) | 13 (13) — grade 1 and 2
renal and urinary disorders (Renal and urinary disorders) | 26 (26) | 42 (42) — grade 1 and 2
reproductive system and breast disorders (Reproductive system and breast disorders) | 19 (19) | 31 (31) — grade 1, 2 and 3
neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4) — grade 2 and 5
respiratory, thoracic and mediastinal disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — grade 1
skin and cubcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) — grade 1
vascular disorders (Vascular disorders) | 8 (8) | 10 (10) — grade 1, 2 and 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-22): https://cdn.clinicaltrials.gov/large-docs/20/NCT03254420/Prot_SAP_000.pdf